CLINICAL TRIAL: NCT04834271
Title: Effects of Blood Flow Restriction Training on Central Mechanisms of Pain Modulation in Subjects With Rotator Cuff Related Shoulder Pain: a Randomized Controlled Trial
Brief Title: Effects of Blood Flow Restriction Training in Rotator Cuff Related Shoulder Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participaints enrolled
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Ruben Fernandez Matias, Clinical Professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020/57
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Subacromial Pain Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise without blood flow restriction (Active Comparator): Side-lying external rotation exercise with a dumbbell (20-30% 1RM) without blood flow restriction.
  Interventions: Other: Side-lying external rotation exercise with a dumbbell
- Exercise with 40% of arterial occlusion pressure blood flow restriction (Experimental): Side-lying external rotation exercise with a dumbbell (20-30% 1RM) with 40% of arterial occlusion pressure blood flow restriction.
  Interventions: Other: Side-lying external rotation exercise with a dumbbell with 40% arterial occlusion pressure blood flow restriction
- Exercise with 80% of arterial occlusion pressure blood flow restriction (Experimental): Side-lying external rotation exercise with a dumbbell (20-30% 1RM) with 80% of arterial occlusion pressure blood flow restriction.
  Interventions: Other: Side-lying external rotation exercise with a dumbbell with 80% arterial occlusion pressure blood flow restriction

INTERVENTIONS:
Other: Side-lying external rotation exercise with a dumbbell — Side-lying external rotation exercise with a dumbbell (20-30% 1RM). 2 times per week during 4 weeks.
  Arms: Exercise without blood flow restriction
Other: Side-lying external rotation exercise with a dumbbell with 40% arterial occlusion pressure blood flow restriction — Side-lying external rotation exercise with a dumbbell (20-30% 1RM) with 40% arterial occlusion pressure blood flow restriction. 2 times per week during 4 weeks.
  Arms: Exercise with 40% of arterial occlusion pressure blood flow restriction
Other: Side-lying external rotation exercise with a dumbbell with 80% arterial occlusion pressure blood flow restriction — Side-lying external rotation exercise with a dumbbell (20-30% 1RM) with 80% arterial occlusion pressure blood flow restriction. 2 times per week during 4 weeks.
  Arms: Exercise with 80% of arterial occlusion pressure blood flow restriction

SUMMARY:
Blood flow restriction training is widespread in sport performance areas, where it has proven to be beneficial in strength and hypertrophy development. However, there are only few studies related to its effects on subjects with pathology, and currently, there is no recent clinical trial evaluating its effects on patients with RCRSP. We are aiming to define the potential benefits, acute and short-term effects of adding blood flow restriction to a low-load exercise training for patients with RCRSP.

ELIGIBILITY:
Inclusion Criteria:

* Pain around the antero-lateral (deltoid area) region of the proximal shoulder during active movements in abduction and/or external rotation.
* 3/5 positive impingement tests: Neer, Hawkins-Kennedy, empty can, painful arc, and resisted external rotation or abduction.
* Pain at rest less than 3cm in a visual analogue scale (VAS).

Exclusion Criteria:

* Previous shoulder surgery.
* Being treated with physical therapy or pharmacogical therapy for shoulder pain.
* External rotation range of motion less than 45º or 50% compared to the contralateral side.
* Suspected shoulder instability (previous dislocation/subluxation, sulcus sign, anterior drawer test, anterior/posterior aprehension test, relocation test).
* Suspected cervical radiculopathy (distraction, spurling, ULNT1, squeeze test, ipsilateral rotation less than 60º)
* Presence of neck pain.
* Suspected rotator cuff tears (drop arm test, external rotation lag sign, diagnostic imaging).
* Contraindications to blood flow restriction therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Conditioned Pain Modulation (CPM) | Baseline, immediately after the first treatment session, 1 month, and 2 months
  Conditioned pain modulation estimated using changes in pressure pain threshold measured with a manual algometer and a sphygmomanometer.

SECONDARY OUTCOMES:
Shoulder pain and disability index (SPADI) | Baseline, 1 month, and 2 months
  The SPADI ranges from 0% (no disability) to 100% (maximum degree of disability)
Pain intensity | Baseline, 1 month, and 2 months
  Mean pain intensity during last week measured with a visual analogue scale (VAS), ranging from 0cm (no pain) to 10cm (worst pain)
Pain-free isometric strength | Baseline, immediately after the first treatment session, 1 month, and 2 months
  Pain-free isometric shoulder external rotation strength measured using a hand-held dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Ruben Fernandez-Matias, Alcalá de Henares, Spain

IPD SHARING:
Plan to Share IPD: No